

## CLINICAL EFFICACY OF BIOMIN F, COLGATE SENSITIVE PRORELIEF AND SENSODYNE RAPID ACTION DENTIFRICES IN DENTIN HYPERSENSITIVITY



SEPTEMBER 7, 2019

NCT04249336

## **CONSENT FORM**

| MR. No Patient name; |
|---|
| Age; Contact number; |
| Address |
| I understand that Drwill use her/his best knowledge, skills and training |
| expertise in my dental examination and treatment of suddenly arising severe pain of short duration |
| in my teeth. I have been fully explained regarding my disease named dentine hypersensitivity, its |
| causes and treatment procedure with potential benefits as |

- Dentine hypersensitivity is a sharp pain of short duration in the teeth due to cold and usually hot drink or food intake. It can be initiated by touch and air blow and vanishes when exposure is removed.
- It occurs by tubular opening in the tooth structure due to either aggressive tooth brushing or wrong tooth brushing technique or excessive use of acidic and carbonated food and drinks.
- I have been informed to refrain from these factors and assured that it can be treated by blocking the openings of tubules with the help of medicinal components present in the toothpaste.
- The Proposed treatment plan is intended to stop severe pain immediately after application of provided tooth paste as well as to prevent the pain arising in future.
- No discomfort is anticipated by application of provided toothpaste.
- I understand that further alternative treatment may be needed later if clinical test of tooth paste doesn't provide intended treatment response.
- Method of proper tooth brushing with the provided tooth paste, brushing time and duration have been explained to me properly.

• My treatment will be done free of cost.

• It is my responsibility to schedule regular dental checkups and follow the instructions of my

doctor regarding treatment method for required treatment response.

Treatment record of the patients will be used for research purpose and for university examination.

I do not have any objection on proposed treatment plan and on sharing my treatment records with

my doctor for this purpose.

\_\_\_\_

Patient's signature